CLINICAL TRIAL: NCT06704945
Title: No Axillary Surgical Treatment in Clinically Lymph Node Negative Patients on Ultrasonography After Neoadjuvant Chemotherapy: A Prospective, Phase III Clinical Trial
Brief Title: No Axillary Surgical Treatment in Clinically Lymph Node Negative Patients on Ultrasonography After Neoadjuvant Chemotherapy
Acronym: Neo-NAUTILUS
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Wonshik Han, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-2410-138-1581
Record Dates: First submitted 2024-11-21; First posted 2024-11-26 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer; Neoadjuvant Therapy; Sentinel Lymph Node Biopsy
Keywords: Omission of axillary surgery after neoadjuvant chemotherapy; Breast cancer; Neoadjuvant chemotherapy; De-escalation; Omission of surgery
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No SLNB group (Experimental): The study arm - BCS without SLNB
  Interventions: Procedure: No axillary surgery
- SLNB group (Other): The control arm - BCS with SLNB(+/-ALND)
  Interventions: Procedure: Axillary surgery

INTERVENTIONS:
Procedure: No axillary surgery — BCS only. Ommission of axillary surgery. No axillary surgery after neoadjuvant chemotherapy.
  Arms: No SLNB group
Procedure: Axillary surgery — BCS with SLNB(+/-ALND)
  Arms: SLNB group

SUMMARY:
NEO-NAUTILUS is a prospective, multicenter, randomized phase III clinical trial to evaluate whether omitting axillary lymph node surgery (ALND or SLNB) in clinically lymph node-negative breast cancer patients after neoadjuvant chemotherapy is non-inferior to performing SLNB in terms of 5-year disease-free survival.

DETAILED DESCRIPTION:
Background:

* No prospective studies have proven that axillary lymph node surgery improves survival in breast cancer patients.
* The ACOSOG Z0011 trial showed that additional axillary dissection did not improve recurrence or survival, even with a 23.7% incidence of non-sentinel node metastases.
* NSABP B-32 established the oncologic safety of SLNB, significantly reducing complications like lymphedema compared to axillary dissection. However, SLNB still carries risks of lymphedema, sensory changes, seromas, and infections.
* The trend has now shifted toward identifying candidates for omitting axillary surgery to minimize unnecessary complications.
* The SOUND trial demonstrated non-inferiority of omitting SLNB in early-stage breast cancer patients with negative axillary ultrasound. Five-year distant metastasis-free survival was comparable between SLNB and no-SLNB groups (97.7% vs. 98.0%).
* Improved ultrasound accuracy (e.g., FNR: 13.7% in SOUND; 11.3% in NAUTILUS) and the therapeutic contribution of whole-breast radiation likely support these findings.
* Patients with a complete pathological response (pCR) in the breast post-NAC rarely have residual lymph node metastases, reducing the need for axillary surgery.
* Single-arm studies (e.g., EUBREAST-01, ASICS, ASLAN) have explored omitting axillary surgery in patients with confirmed breast pCR. However, these studies face limitations due to small sample sizes, single-arm design, and the necessity of axillary surgery if pCR is not achieved.
* To address these limitations, the NEO-NAUTILUS trial proposes the first randomized trial to compare disease-free survival and local recurrence rates between patients who omit SLNB (experimental group) and those who undergo SLNB (control group) after NAC, focusing on patients deemed axillary node-negative by ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Women aged ≥19 years.
* Histologically confirmed invasive breast carcinoma treated with neoadjuvant chemotherapy.
* Clinical staging prior to NAC: cT1-3, cN0, M0 (AJCC 8th Edition).
* If pre-NAC staging is cT1-3, cN1, M0, must meet the following criteria:

  1. HER2-positive or triple-negative breast cancer (TNBC).
  2. At least 30% reduction in tumor size on MRI after NAC (comparing pre- and post-NAC MRI).
* Negative axillary lymph node status on ultrasound after NAC.
* Planned for breast-conserving surgery with completed neoadjuvant chemotherapy (at least half the planned regimen must be completed).
* ECOG performance status of 0-2.
* Signed written informed consent before enrollment.

Exclusion Criteria:

* History of any cancer within the past 5 years.
* Bilateral breast cancer.
* Patients requiring mastectomy.
* Tumor size >5 cm after NAC.
* Male breast cancer.
* Pregnant or breastfeeding women.
* Inability to understand and complete questionnaires.

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 464 (Estimated)
Dates: Start 2025-06-04 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2034-12-31 (Estimated)

PRIMARY OUTCOMES:
Invasive Disease Free Survival (iDFS) | 5 years
  Evaluate invasive disease free survivals

SECONDARY OUTCOMES:
Overall Survival (OS) | 5 years
  Evaluate overall survival
Distant Metastasis Free Survival (DMFS) | 5 years
  Evaluate distant metastasis free survival
Axillary recurrence rate | 5 years
  Evaluate ipsilateral axillary recurrence rate
Locoregional Recurrence Rate (LRR) | 5 years
  Evaluate locoregional recurrence rate
QoL | 1 year
  Evaluate Quality of Life of patient by EORTC QLQ-C30 questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hopsital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes
Study protocol will be shared.
Supporting Information: Study Protocol
Time Frame: The study protocol will be published as a journal article.
Access Criteria: Anyone interested in viewing the study protocol will be able to access it through the published journal.

REFERENCES:
- [Background] Jung JG, Ahn SH, Lee S, Kim EK, Ryu JM, Park S, Lim W, Jung YS, Chung IY, Jeong J, Chang JH, Shin KH, Chang JM, Moon WK, Han W. No axillary surgical treatment for lymph node-negative patients after ultra-sonography [NAUTILUS]: protocol of a prospective randomized clinical trial. BMC Cancer. 2022 Feb 20;22(1):189. doi: 10.1186/s12885-022-09273-1. PMID 35184724
- [Derived] Jung JJ, Kim HJ, Chae BJ, Kim EK, Ahn JH, Jeong J, Lee S, Jung SP, Woo J, Min J, Cheun JH, Chung MS, Shin KH, Chang JM, Moon WK, Han W. A Randomized Trial of Sentinel Node Biopsy Omission After Neoadjuvant Systemic Therapy in Clinically Node-Negative or Selected Node-Positive Breast Cancer. J Breast Cancer. 2025 Dec;28(6):437-447. doi: 10.4048/jbc.2025.0157. Epub 2025 Nov 14. PMID 41311332